CLINICAL TRIAL: NCT02102698
Title: Ecopipam Treatment of Tourette's Syndrome in Subjects 7-17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSY302
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2016-11

CONDITIONS: Tourette's Syndrome
Keywords: Tourette's Syndrome; Ecopipam; D1 Receptor; Phase 2
MeSH Terms: conditions — Tourette Syndrome | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ecopipam (Experimental): Ecopipam is a selective antagonist of the dopamine D1/D5 receptor family that is being studied as a treatment for Tourette's Syndrome
  Interventions: Drug: Ecopipam
- Placebo (Placebo Comparator): Placebo is the inactive comparator
  Interventions: Drug: Ecopipam

INTERVENTIONS:
Drug: Ecopipam — Ecopipam is a selective antagonist of the dopamine D1 receptor family.
  Other Names: SCH 39166; PSYRX101

SUMMARY:
Tourette's Syndrome is a neurological disease characterized by motor and vocal tics. It has been hypothesized that abnormal interactions of dopamine with its receptors may cause the tics. The purpose of this study is to test the hypothesis that a drug (ecopipam) that selectively blocks dopamine D1/D5 receptors can reduce the frequency and severity of the tics.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled crossover study to determine whether ecopipam can reduce the symptoms of Tourette's in children age 7-17 years.

ELIGIBILITY:
Inclusion Criteria:• Subjects must have Tourette's Syndrome (TS) based on the clinician-administered Diagnostic Confidence Index (DCI) for TS.

* Subjects must exhibit both motor and vocal tics.
* Subjects must have a minimum score of 20 at both Screening and Baseline (just prior to the first treatment) on the Yale Global Tic Severity Scale.
* Subjects must be age (≥ 7 to < 18 years of age)
* Subjects must weigh ≥ 20 kg (45 lbs)
* Adolescent females of childbearing potential who are sexually active must be using effective contraception (i.e., oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for the duration of their participation in the study. They must also agree to use contraception for 30 days after their last dose of study drug.
* Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.
* Subject's parent or legal guardian must execute a written informed consent.
* Subject must execute a written informed assent.

Exclusion Criteria:

* Subjects who have unstable medical illness or clinically significant abnormalities on laboratory tests, or ECG at Screening.
* Subjects with a major depressive episode in the past 2 years
* Subjects with a history of attempted suicide
* Subjects with clinically significant suicidality (based on the Columbia Suicide Rating Scale (C-SSRS)
* Subjects with a first-degree relative with a major depressive episode that resulted in any psychiatric hospitalization, or attempted/ completed suicide with the exception of a hospitalization for post-partum depression.
* Subjects with a history of seizures (excluding febrile seizures that occurred >2 years in the past)
* Subjects with a myocardial infarction within 6 months.
* Girls who are currently pregnant or lactating.
* Subjects who have a need for medication (other than ecopipam) with possible effects on TS symptoms (i.e., lithium, psychostimulants)
* Subjects who have a need for medications which would have unfavorable interactions with ecopipam, e.g., dopamine antagonists or agonists [including bupropion], tetrabenazine, or monoamine oxidase inhibitors.
* Subjects with a lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any psychotic disorder determined by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders - 4th Edition (DSM-IV) Axis-I Disorders (SCID).
* Subjects with current or recent (past 3 months) DSM-IV substance abuse or dependence (with the exception of nicotine).
* Subjects with positive urine drug screen (cocaine, amphetamine, methamphetamine, tetrahydrocannabinol (THC), benzodiazepines, barbiturates, phencyclidine (PCP), opiates) at Screening. Subjects with urine positive only for benzodiazepines and/or marijuana (i.e., a user but not an abuser as based on DSM-IV criteria) may be eligible.
* Subjects who have had previous treatment with ecopipam.
* Subjects who have had treatment with:

  * investigational medication within 3 months of starting study
  * depot neuroleptics within 3 months of starting study
  * other psychotropics with possible effects on TS symptoms (i.e., lithium, tetrabenazine) within 2 weeks prior to Screening.
  * oral neuroleptics within 4 weeks
  * selective serotonin reuptake inhibitors unless the dosage has been stable for a minimum of 4 weeks prior to study start and not prescribed to relieve the neurological signs of TS

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale | 30 days
  The Yale Global Tic Severity Scale (YGTSS) is the standard rating scale used to assess the effects of a new treatment on the symptoms of Tourette's Syndrome.

SECONDARY OUTCOMES:
Adverse events (SAE), clinical laboratory values, regular measurement of vital signs, electrocardiograms, C-SSRS, Children's Depression Inventory and Physical Exams. | 30 days
  Safety evaluations are included.
DuPaul ADHD rating scale-IV | 30 days
  This is a validated rating scale for the symptoms of attention deficit disorder. This is included because people with Tourette's often have attention deficit hyperactivity disorder (ADHD) as well.
Child Yale-Brown Obsessive Compulsive Scale | 30 days
  This is validated rating scale which measures symptoms of obsessive-compulsive behaviors. People with Tourette's often also show symptoms of obsessive-compulsive behaviors.
Children's Depression Inventory | 30 days
  The Children's Depression Inventory is a validate rating scale which measures signs of depression of in children. People with Tourette's often report feelings of depression. In addition, treatment with ecopipam has been reported to increase signs of depression in some patients.
Clinical Global Impression - Improvement and Severity Scales | 30 days
  Clinical Global Impression Scales (improvement and severity) are validated rating scales that measure whether the treatment improves the symptoms of the disease (CGI-I) and whether the treatment reduces the severity of the disease (CGI-S)
Columbia-Suicide Severity Rating Scale | 30 days
  The Columbia Suicide Severity Rating Scale is a validated rating scale which measures feelings of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Gilbert, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (11):
- United States (11):
  - UCLA, Los Angeles, California
  - University of South Florida/Rothman Center for Neuropsychiatry, St. Petersburg, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - University of Chicago Medical School, Chicago, Illinois
  - Children's Mercy Kansas City, Kansas City, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Overlook Hospital, Summit, New Jersey
  - North Shore-Long Island Jewish Hosptial, Manhasset, New York
  - Weill Cornell Medical School, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Gilbert DL, Budman CL, Singer HS, Kurlan R, Chipkin RE. A D1 receptor antagonist, ecopipam, for treatment of tics in Tourette syndrome. Clin Neuropharmacol. 2014 Jan-Feb;37(1):26-30. doi: 10.1097/WNF.0000000000000017. PMID 24434529
- [Derived] Gilbert DL, Murphy TK, Jankovic J, Budman CL, Black KJ, Kurlan RM, Coffman KA, McCracken JT, Juncos J, Grant JE, Chipkin RE. Ecopipam, a D1 receptor antagonist, for treatment of tourette syndrome in children: A randomized, placebo-controlled crossover study. Mov Disord. 2018 Aug;33(8):1272-1280. doi: 10.1002/mds.27457. Epub 2018 Sep 7. PMID 30192018